CLINICAL TRIAL: NCT06269302
Title: Comparison of the Effect of Warfarin and Direct Oral Anticoagulants on Upper Gastrointestinal System Bleeding
Brief Title: Comparison of the Effect of Warfarin and Direct Oral Anticoagulants
Status: Completed | Type: Observational
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Duriye Sila Karagoz Ozen, MD, Internal Medicine Specialist, Samsun Education and Research Hospital
Other Study IDs: 2
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Anticoagulants and Bleeding Disorders; Gastrointestinal Hemorrhage
Keywords: Gastrointestinal System; Oral Anticoagulant; Rebleeding; upper gastrointestinal system bleeding
MeSH Terms: conditions — Hemostatic Disorders; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with recurrent gastrointestinal bleeding: The data of all patients who applied to Samsun Training and Research Hospital for 12 months in 2022 and diagnosis of upper gastrointestinal bleeding and hospitalized by Internal Medicine and Gastroenterology clinics or who underwent outpatient endoscopy were included in the study.Patients who had recurrent upper GI bleeding were detected by controlling them over the hospital software system and by reaching each patient again. The frequency of use of new generation oral anticoagulants in patients with rebleeding was determined, and data such as rebleeding rate, length of hospital stay, need for transfusion, and mortality were analyzed in the groups who did not use this drug and those who used it.

SUMMARY:
In this study, it was aimed to compare the frequency of new oral anticoagulants and warfarin usage, and to reveal the rates of recurrent upper gastrointestinal bleeding among patients who applied to our hospital with upper gastrointestinal bleeding

DETAILED DESCRIPTION:
The data of all patients who applied to Samsun Training and Research Hospital Internal Medicine with a diagnosis of upper gastrointestinal bleeding and hospitalized by Internal Medicine and Gastroenterology clinics or who underwent outpatient endoscopy between 01.01.2021 and 31.12.2021 were included. The patients' data were analyzed from the patient files and hospital automation system retrospectively. Patients who had recurrent upper GI bleeding were detected by controlling them over the hospital software system and by reaching each patient again. The frequency of the new generation oral anticoagulants usage in patients with re-bleeding was determined, and data such as re-bleeding rate, length of hospital stay, need for transfusion, and mortality were analyzed in the groups who did not use this drug and those who used it. The patient demographics were also compared between the groups who were using the new generation oral anticoagulants, acetylsalicylic acid or warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Upper gastrointestinal bleeding
* 12 months follow-up

Exclusion Criteria:

* Age <18 years old
* Lower gastrointestinal bleeding
* Esophageal variceal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were admitted to Samsun Training and Research Hospital with a diagnosis of upper gastrointestinal bleeding and hospitalized by Internal Medicine and Gastroenterology clinics or who underwent outpatient endoscopy were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the incidence of recurrent bleeding | 12 months
  Increase or decrease in the incidence of recurrent bleeding

CONTACTS AND LOCATIONS:
Overall Officials: DÜRİYE SILA KARAGÖZ ÖZEN, MD, Principal Investigator — Samsun Education and Research Hospital
Locations (1):
- Samsun Education and Research Hospital, Samsun, İlkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided